CLINICAL TRIAL: NCT05849207
Title: IIT2022-03-Paquette-GeriBMT: A Phase I Study of De-Escalation of Post-Transplant Cyclophosphamide Dosing in Patients Aged >/= 65 Years Undergoing Conditioning With Fludarabine and Total Body Irradiation 800 cGy
Brief Title: Post-Transplant Cyclophosphamide in Patients Aged >/= 65 Years Undergoing Haploidentical Transplant
Acronym: GeriBMT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ronald Paquette (Other)
Responsible Party: Sponsor-Investigator, Ronald Paquette, Medical Director, Blood and Marrow Transplant Program, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022-03-PAQUETTE-GERIBMT
Record Dates: First submitted 2023-04-13; First posted 2023-05-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Hematologic Malignancies
Keywords: Allogeneic Transplantation
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Open-label trial
  De-escalation of post-transplant cyclophosphamide dosing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Arm (Experimental): All patients will receive cyclophosphamide on Day +3 and Day +4 following transplant.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide will be administered at 50, 40, 32, or 25 mg/k/d intravenous infusion (IV) continuously for two days starting 60-72 hours after transplant.

SUMMARY:
The purpose of this phase 1 study is to determine the optimal dose of the immune suppressive drug, cyclophosphamide, following standard allogeneic stem cell transplant in patients aged >/= 65 years with hematologic malignancies.

DETAILED DESCRIPTION:
The patients will receive a standard dose, or a reduced amount of the immune suppressive drug, cyclophosphamide, that is routinely administered after the transplant procedure. The following procedures will be performed: cardiac MRI scans and/or transthoracic echocardiogram (TTE); laboratory tests, geriatric assessments and tests to measure strength and stability.

Participation in the study is expected to last up to one year with follow-up visits occurring on Day +30, Day +100, Day +180 and Day +365 following allogenic stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >/= 65 years
* Patient and related Donor (if applicable) sign the Informed Consent Form for the study. If donor is unrelated, donor does not sign Informed Consent Form and this will not affect recipient study eligibility.
* Patient meets standard criteria for allogeneic stem cell transplant
* Patient is deemed suitable to receive Flu/TBI 800 conditioning regimen as standard of care transplant
* Donor is willing to donate peripheral blood stem cells

Exclusion Criteria:

* Patient has a diagnosis of myelofibrosis
* Patient has high titer antibodies (>10,000 mean fluorescent intensity) against one or more donor HLA antigens
* Patient has undergone prior autologous or allogeneic stem cell transplant
* Requiring sedation for cardiac MRIs.
* Prohibited Implants and/or Devices:

  * Mechanical, magnetic or electrical activated implants (i.e. cardiac pacemakers, neurostimulators and infusion pumps)
  * Ferromagnetic implants and ferromagnetic foreign bodies, such as intracranial, aneurysm clips, shrapnel and intraocular metal chips as these could become dislodged.
* Subjects with claustrophobia, problems being in enclosed spaces, or inability to lie supine.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximum grade acute GVHD by day +100 by Modified Keystone Criteria | 100 days post-transplant
  Evaluate the frequency of grade III/IV acute GVHD using Modified Keystone Criteria

SECONDARY OUTCOMES:
Time to neutrophil and platelet engraftment | 60 days post-transplant
  Days to neutrophil and platelet engraftment since transplant
Non-Relapse mortality | 100 days post-transplant
  Rate of treatment-related mortality
Chronic Graft Versus Host Disease (GVHD) at 1 year | 1-year post-transplant
  * Rate and severity of patients with chronic GVHD at day 365 post-transplantation.
  * Chronic GVHD is when the donated stem cells attack the body after 100 days post-transplant. Chronic GVHD is defined by NIH Consensus Criteria for chronic GVHD.
Relapse | 1-year post-transplant
  Percentage of patients who relapse by year 1
Overall Survival (OS) | 1-year post-transplant
  Overall survival at 1 year
Graft Versus Host Disease (GVHD)-free and Relapse Free Survival | 1-year post- transplant
  Percentage of patients without relapse or GVHD at 1 year
Change in cardiac function | From 60 days prior to transplant to 365 days post-transplant
  Change in cardiac (heart) injury defined by any of an increase in T1 time > 500 ms from pre-transplant imaging, T2 time > 5 ms from pre-transplant imaging, or a decrease in left ventricular ejection fraction > 10% of the original measurement to below 53% from post-transplant imaging.
Change in active daily living | From 60 days prior to transplant to 365 days post-transplant
  Change in function over time as determined by Lawton Activities of Daily Living questionnaire.
  - Patients will choose either 0 or 1 to rate their level of function with 1 being the highest level of function.
Change in function | From 60 days prior to transplant to 365 days post-transplant
  Change in function over time as determined by the Patient-Reported Outcomes Measurement Information System (PROMIS) Cancer Function Brief 3-Dimensional Profile.
  - Patients will rate their physical condition and fatigue using an inverse 5-item likert scale where 5 represents the highest level of function or the greatest amount of impact on function.
Change in pain | From 60 days prior to transplant to 365 days post-transplant
  Change in pain over time as determined by the Patient-Reported Outcomes Measurement Information System (PROMIS) Cancer Function Brief 3-Dimensional Profile.
  - Patients will rate their level of pain using a scale from 0 to 10 with 10 being the highest level of pain.
Change in physical function | From 60 days prior to transplant to 365 days post-transplant
  Change in lower limb functioning over time as evaluated by the Short Physical performance Battery. (SPPB).
  - Patients will complete a series of tests evaluating balance, speed and standing capabilities. Patients will be rated using a scale of 0 to 12 where a score of less than 10 indicates mobility limitations.
Change in grip strength | From 60 days prior to transplant to 365 days post-transplant
  Change in grip strength as measured using the Jamar dynamometer (device used to measure grip)
Change in cognitive function | From 60 days prior to transplant to 365 days post-transplant
  Change in cognitive function over time using the Patient-Reported Outcomes Measurement Information System (PROMIS) Cognition questionnaire.
  -Patients will rate their cognitive ability on a scale of 1 to 5 with 5 representing the least amount of difficulty.
Change in mental health | From 60 days prior to transplant to 365 days post-transplant
  Change in mental health over time using the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 Depression Questionnaire.
  - Patients will rate their level of depression on a scale of 1 to 5 with 5 representing the greatest level of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Paquette, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No